CLINICAL TRIAL: NCT03159221
Title: Behavioral Family Systems Therapy for Teens With Type 2 Diabetes: A Pilot
Brief Title: Behavioral Family Systems Therapy (BFST) for Teens With Type 2 Diabetes
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Lisa Buckloh, PhD, Clinical Research Psychologist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Buckloh
Record Dates: First submitted 2015-10-06; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2; Childhood Obesity
Keywords: type 2 diabetes in adolescents; obesity in adolescents; behavioral family systems therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BFST for Teens with Type 2 Diabetes (Experimental): Psychological intervention: Families randomized to the intervention group will receive 12 sessions of Behavioral Family Systems Therapy for Teens with type 2 diabetes (BFST-DM2) over 6 months.
  Interventions: Behavioral: BFST for Teens with Type 2 Diabetes
- Control group (Standard Care) (No Intervention): The participants assigned to the control group will receive their standard medical care for diabetes.

INTERVENTIONS:
Behavioral: BFST for Teens with Type 2 Diabetes — BFST for Teens with Type 2 Diabetes: 12 (90 minute sessions) over 6 months of Behavioral Family Systems Therapy (BFST), delivered by a Licensed clinical social worker. BFST consists of 4 components: problem-solving, communication skills training, cognitive restructuring, and functional and structural family therapy.
  Other Names: BFST - Behavioral Family Systems Therapy
  Arms: BFST for Teens with Type 2 Diabetes

SUMMARY:
This is a randomized, controlled pilot trial of Behavioral Family Systems Therapy for Teens with Type 2 Diabetes (BFST-DM2), an individual psychological intervention tailored to meet the needs of teens with type 2 diabetes. It is hypothesized that this behavioral family intervention will be feasible to implement with teens with type 2 diabetes and will have positive effects on treatment adherence, health outcomes like weight status and metabolic control, and psychological outcomes.

DETAILED DESCRIPTION:
The incidence of type 2 diabetes mellitus (DM2) in youth is increasing dramatically with the rise in obesity in the U.S. and worldwide. DM2 in youth, as with adults, is clearly linked to modifiable risk factors such as obesity, sedentary lifestyle, and poor diet. Youth with DM2 are at increased risk for medical complications such as cardiovascular disease, retinopathy, and neuropathy, as well as psychological problems such as depression, anxiety, poor self-esteem, eating disorders, and poor coping and problem solving. Although there are studies demonstrating that family-based lifestyle and psychological interventions are successful in reducing obesity in youth and in improving metabolic control and adherence in youth with type 1 diabetes mellitus (DM1), very little has been published on potential lifestyle or psychological treatments for youth with DM2. Studies have shown that Behavioral Family Systems Therapy (BFST) has been effective in improving metabolic control, adherence, family communication, and problem solving in youth with DM1. This intervention could be effective in treating youth with DM2, as many of the skills necessary for good metabolic control, health outcomes, treatment adherence, and psychological adjustment are similar in both populations. This application proposes a randomized, controlled pilot trial of BFST-DM2, an individual psychological intervention tailored to meet the needs of teens with DM2. BFST will be adapted to make this intervention more feasible and relevant with minority and low-income populations and also to focus on weight management, exercise, and nutrition. The BFST-DM2 intervention includes 12 (90-minute) sessions over 6 months. Areas targeted for improvement will include metabolic control, weight/body mass index, treatment adherence, family lifestyle choices (activity, diet), family communication, and problem solving. One of the main aims of this pilot study is to gather exploratory information on the effectiveness of the BFST-DM2 intervention on measures of health outcomes, medical adherence, lifestyle changes, and family problem-solving and communication skills. In addition, it is an aim to estimate treatment effect size to determine the sample size needed to power a larger multi-site trial of the BFST-DM2 intervention. Other aims include determining factors associated with feasibility (recruitment, retention, participation, generalizability) as well as to modify the intervention to be culturally sensitive and to be more relevant to the individual needs of the DM2 adolescent population. The BFST-DM2 intervention will be compared with standard medical therapy on measures of health outcomes (metabolic control, body mass index, weight, waist circumference, body fat) physical activity (accelerometer), nutritional intake, treatment adherence, psychological adjustment (self-esteem, quality of life), family communication, and problem solving. The researchers will analyze predictors of treatment outcome and the treatment effects at the immediate post-treatment interval (6 months from baseline). Health outcomes and medical adherence data also will be collected 12 months from baseline to determine maintenance of treatment effects over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus for 6 months or more
* Age-adjusted Body Mass Index at or above the 85th percentile (considered overweight)
* Established diabetes care in Nemours Children's Clinic system or diabetes care meets minimum criteria for current American Diabetes Association Standards.
* Adolescent lives at home in the study geographical area (Jacksonville, FL)over the course of the study duration (one year).
* One caregiver in the home is willing to participate in the family intervention.

Exclusion Criteria:

* Adolescent has another systemic chronic disease other than well-controlled asthma.
* Genetic syndrome or disorder (other than diabetes) known to affect glucose tolerance.
* Daily use of glucocorticoids or other medications known to affect glucose tolerance.
* Teen is enrolled in special education for students who have autism or are mentally handicapped.
* Adolescent is pregnant or planning to be pregnant within 1 year.
* Teen resides in temporary foster care, group home, or juvenile detention center.
* The family has an open case with an agency investigating child abuse or neglect.
* Adolescent has been in an inpatient psychiatric facility or substance abuse treatment in the past 6 months.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (weight status) at 6 months and at 12 months | baseline, 6 months after baseline, 12 months after baseline
  Body Mass Index (adjusted for height, gender, and age) - height and weight in kg and meters (kg/m^2) - change in BMI across time points is being studied - change in weight from baseline to 6 months and change in weight from baseline to 12 months

SECONDARY OUTCOMES:
metabolic control (HbA1c) | baseline, 6 months after baseline, 12 months after baseline
  Metabolic control is measured using HbA1c values
Treatment Adherence | baseline, 6 months after baseline, 12 months after baseline
  Treatment Adherence is measured using the Diabetes Self Management Survey for Teens with Type 2 Diabetes.
Family Problem-solving | baseline, 6 month after baseline
  Family problem-solving is measured using the Revised Diabetes Family Conflict Scale
Physical activity | baseline, 6 months after baseline
  Physical activity is measured by an accelerometer
Body Fat (weight status) | baseline, 6 months after baseline, 12 months after baseline
  Body fat percent change - measured by a hand-held body fat impedance device
Waist Circumference (weight status) | baseline, 6 months after baseline, 12 months after baseline
  Waist circumference in cm
Food intake | baseline, 6 months after baseline
  Nutrition/food intake as measured by the Nutrition Data Systems for Research interview
Family communication skills | baseline, 6 months after baseline
  Family communication skills are measured by the Family Communication (Interaction Behavior Code)
Teen Self-esteem | baseline, 6 months after baseline
  Teen Self-Perception/Self-esteem is measured by the Harter Self-Perception Profile
Teen Quality of Life | baseline, 6 months after baseline
  Teen Quality of Life is measured by The Pediatric Quality of Life Inventory (PedsQL)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Buckloh, Ph.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Specialty Care, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No